CLINICAL TRIAL: NCT02764866
Title: Prevalence of Sleep Apnea in Lung Cancer
Brief Title: Sleep Apnea in Lung Cancer: A Prospective Study
Acronym: SAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, LUIS SEIJO MACEIRAS, Attending physician, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: InstitutoFJD
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer; Sleep-Disordered Breathing
Keywords: Lung cancer; Sleep apnea; Sleep disordered breathing
MeSH Terms: conditions — Lung Neoplasms; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleep testing (Experimental): Enrolled patients with lung cáncer will undergo home sleep testing during their initial oncologic evaluation, prior to treatment.
  Interventions: Other: Sleep testing

INTERVENTIONS:
Other: Sleep testing — Home sleep testing

SUMMARY:
The study seeks to determine the prevalence of sleep disordered breathing in a population of patients diagnosed with lung cáncer.

DETAILED DESCRIPTION:
Obstructive sleep apnea hypopnea syndrome (OSAHS) is an important medical condition which causes significant morbidity and mortality. The prevalence of OSAHS in Spain is 4-6% in men and 2-4% in women and rises steadily with age. Snoring and smoking have been independently linked, and smoking may be a risk factor for developing OSAHS. This is particularly true of heavy smokers (> 2 packs/day), those at greatest risk for LC. Associations between OSAHS and some forms of cancer have been described in humans, especially in those experiencing nocturnal hypoxemia, and intermittent hypoxia has been linked to the progression of cancer in animal models. LC is currently the leading cause of cancer deaths in developped nations. A link between OSAHS and LC, therefore, is plausible.

Sleep disordered breathing may be common among patients recently diagnosed of lung cancer and may contribute to tumor progression.

Objectives: a) To perform home sleep testing in patients recently diagnosed with lung cancer in order to determine the prevalence of sleep disordered breathing in this patient population. b) To include biological samples obtained from all participants, including surgically treated patients with stage I / IIp LC through the program in the CIBERES Pulmonary Biobank Platform. Biological samples will be preserved under different storage conditions for subsequent determination of molecular biomarkers. c) To follow-up lung cancer patients with and without sleep disordered breathing in order to determine the potential influence OSAHS might have on their prognosis.

Prospective screening for sleep disordered breathing will be performed by home sleep testing in 100 subjects diagnosed with lung cancer, irrespective of stage at diagnosis, who give their consent. A modified epidemiologic questionnaire for sleep disordered breathing will also be administered. Patients identified as suffering from OSAHS will be referred to sleep clinic. Biologic samples and lung function studies will be obtained in all participating patients.

All patients with lung cancer will undergo follow-up for at least three years or until their demise, and those identified with OSAHS will also be followed in sleep clinic. The prevalence of OSAHS in this patient population will be determined. A link between OSAHS, and especially intermittent nocturnal hypoxemia, and tumor progression will be sought.

ELIGIBILITY:
Inclusion Criteria:

* All patients with recently diagnosed lung cancer, inlcuding all stages of disease.

Exclusion Criteria:

* Patients unable to comply with home sleep testing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-02; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of sleep disordered breathing in lung cancer | 12 months

SECONDARY OUTCOMES:
Survival of lung cancer in patients with sleep disordered breathing | 36 months
Lung cancer stage in patients with sleep disordered breathing | 12 months
Lung cancer progression free survival in patients with sleep disordered breathing | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Seijo, MD, PhD, Principal Investigator — Instituto de Investigacion Fundacion Jimenez Diaz
Locations (1):
- Fundacion Jimenez Diaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Seijo LM, Perez-Warnisher MT, Giraldo-Cadavid LF, Oliveros H, Cabezas E, Troncoso MF, Gomez T, Melchor R, Pinillos EJ, El Hachem A, Gotera C, Rodriguez P, Gonzalez-Mangado N, Peces-Barba G. Obstructive sleep apnea and nocturnal hypoxemia are associated with an increased risk of lung cancer. Sleep Med. 2019 Nov;63:41-45. doi: 10.1016/j.sleep.2019.05.011. Epub 2019 Jun 6. PMID 31605903
- See also: Lung cancer screening home web page — http://www.lungscreen.eu